CLINICAL TRIAL: NCT01446003
Title: A Multiple-Dose Clinical Trial to Study the Effect of MK-8457 on Ambulatory Blood Pressure in Hypertensive Patients
Brief Title: A Study of the Effect of MK-8457 on Blood Pressure in Hypertensive Participants (MK-8457-004-AM1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 8457-004
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-8457-Placebo Sequence (Experimental): Participants received MK-8457 100 mg twice daily (BID) for 10 days followed by Placebo for 10 days. Each treatment was separated by a 10-day washout.
  Interventions: Drug: MK-8457; Drug: Placebo for MK-8457
- Placebo-MK-8457 Sequence (Experimental): Participants received Placebo for 10 days followed by MK-8457 100 mg BID for 10 days. Each treatment was separated by a 10-day washout.
  Interventions: Drug: MK-8457; Drug: Placebo for MK-8457

INTERVENTIONS:
Drug: MK-8457 — 10 x 10-mg capsule BID for 10 days
Drug: Placebo for MK-8457 — 10 x 10-mg capsule BID for 10 days

SUMMARY:
This study will evaluate the effect of treatment with multiple doses of MK-8457 on systolic blood pressure in participants with mild to moderate hypertension in addition to safety and tolerability. The study hypothesis is that MK-8457 does not increase systolic blood pressure to a clinically significant extent, as measured by 24-hour mean ambulatory systolic blood pressure change from baseline after 10 days of dosing.

ELIGIBILITY:
Inclusion Criteria:

* If female, must be of non-childbearing potential
* If male with female partner(s) of child-bearing potential must agree to use a medically acceptable method of contraception during the study and for 90 days after the last dose of study drug
* Body mass index (BMI) ≤35 kg/m^2
* Mild-to-moderate hypertension requiring treatment with one or more antihypertensive agents
* Receiving stable treatment for hypertension for at least 8 weeks prior to the start of dosing and continuing therapy for duration of study
* No clinically significant arrhythmias or clinically significant abnormality on electrocardiogram
* Nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months

Exclusion Criteria:

* Any illness that might confound the results of the study or poses an additional risk
* History of stroke, chronic seizures, or major neurological disorder
* Clinically significant endocrine, gastrointestinal, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Clinically significant cardiovascular disease or has active angina
* History of malignant neoplastic disease
* Taking 325 mg aspirin daily
* Taking 3 or more medications for the treatment of hypertension
* Unable to refrain from or anticipates the use of any non-steroidal anti-inflammatory drugs (NSAIDs)
* Consumes excessive amounts of alcohol and/or coffee, tea, cola, or other caffeinated beverages
* Has had major surgery, donated or lost 1 unit of blood or participated in another investigational study within 4 weeks
* Significant multiple and/or severe allergies
* Regular user of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10-25 (Actual); Primary Completion 2012-02-18 (Actual); Study Completion 2012-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Call for Information, Miramar, Florida
  - Call for Information, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | MK-8457-Placebo Sequence | Placebo-MK-8457 Sequence
Started | 16 | 15
Completed | 14 | 15
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0
Period: Period 2
Arm/Group | MK-8457-Placebo Sequence | Placebo-MK-8457 Sequence
Started | 14 | 15
Completed | 13 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants that received treatment with either MK-8457 or Placebo in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (5.9)
Age, Customized [Number; unit: Participants]
  Between 18 and 65 years | 30
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 10 in 24-hour Mean Ambulatory Systolic Blood Pressure (SBP)
Description: SBP was measured using ambulatory blood pressure monitoring (ABPM) on Day -1 and Day 10 of each treatment period. The 24-hour least squares (LS) mean ambulatory SBP change from baseline was then determined for Day 10, the last day of multiple dose treatment. Baseline is defined as the average 24-hour SBP for each participant on Day -1. Increased values represent an increase in hypertensive severity.
Time Frame: Baseline and Day 10
Population: The per-protocol population consisting of participants who comply with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment according to the underlying scientific model used for analysis (change in 24-hour mean ambulatory SBP).
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- MK-8457 100 mg BID: Participants received MK-8457 100 mg BID for 10 days followed by Placebo for 10 days. Each treatment was separated by a 10-day washout.
- Placebo: Participants received Placebo for 10 days followed by MK-8457 100 mg BID for 10 days. Each treatment was separated by a 10-day washout.
Arm/Group | MK-8457 100 mg BID | Placebo
Number analyzed (Participants) | 29 | 28
mmHg | -0.47 [-2.60 to 1.66] | -2.49 [-4.66 to -0.31]
Statistical Analysis 1: Comparison: MK-8457 100 mg BID vs Placebo; If the upper limit of the 90% confidence interval lies below the bound 5 mmHg, the hypothesis that change from baseline in ambulatory 24-hour mean SBP in participants with mild to moderate hypertension following 10 days of multiple dosing of MK-8457 is similar to placebo will be supported; Test type: Superiority or Other; Linear mixed effect models; The model contained period and treatment as fixed effect, Day -1 baseline as a fixed continuous covariate, and participant as random effect; Mean Difference (Final Values) = 2.02, 90% CI 2-sided [-0.52 to 4.56]

2. Secondary Outcome: Change From Baseline to Day 10 in 24-hour Mean Ambulatory Diastolic Blood Pressure (DBP)
Description: DBP was measured using ambulatory blood pressure monitoring (ABPM) on Day -1 and Day 10 of each treatment period. The 24-hour LS mean ambulatory DBP change from baseline was then determined for Day 10, the last day of multiple dose treatment. Baseline is defined as the average 24-hour DBP for each participant on Day -1. Increased values represent an increase in hypertensive severity.
Time Frame: Baseline and Day 10
Population: The per-protocol population consisting of participants who comply with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment according to the underlying scientific model used for analysis (change in 24-hour mean ambulatory DBP).
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | MK-8457 100 mg BID | Placebo
Number analyzed (Participants) | 29 | 28
mmHg | 0.22 [-1.33 to 1.78] | -1.35 [-2.93 to 0.23]
Statistical Analysis 1: Comparison: MK-8457 100 mg BID vs Placebo; Test type: Superiority or Other; Linear mixed effects model; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 1.57, 90% CI 2-sided [0.19 to 2.96]

3. Secondary Outcome: Change From Baseline to Day 10 in Maximum Moving Average (maxMAΔ) Blood Pressure Measured Over 4 Hours
Description: The effect of drug on resting blood pressure was estimated using maxMAΔ. The maxMAΔ in blood pressure was calculated as the maximum moving average change from baseline to Day 10 of 3 consecutive 15-minute blood pressure measurements across the first 4 hours after the morning (AM) and evening (PM) doses. In this method, the LS means of three consecutive time points over the 4 hour period were determined and the maximum LS mean was used for the endpoint. Blood pressure was determined using continuous monitoring at rest. Increased values represent an increase in hypertensive severity.
Time Frame: Up to 4 hours postdose on Days 1 and 10
Population: The per-protocol population consisting of participants who comply with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment according to the underlying scientific model used for analysis (maxMAΔ in blood pressure).
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | MK-8457 100 mg BID | Placebo
Number analyzed (Participants) | 29 | 28
mmHg
  SBP - AM (n=29,28) | 17.80 (13.36) [12.36 to 23.23] | 9.90 (10.05) [4.37 to 15.43]
  SBP - PM (n=29,27) | 12.68 (12.28) [8.63 to 16.72] | 13.61 (11.31) [9.40 to 17.83]
  DBP - AM (n=29,28) | 16.90 (8.17) [13.14 to 20.66] | 11.64 (8.26) [7.80 to 15.48]
  DBP - PM (n=29,27) | 10.89 (11.52) [8.02 to 13.76] | 12.58 (10.89) [9.60 to 15.56]
Statistical Analysis 1: Comparison: MK-8457 100 mg BID vs Placebo; Treatment comparison of maxMAΔ in SBP from baseline to Day 10 after AM dosing; Test type: Superiority or Other; Linear mixed effects model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.90, 90% CI 2-sided [2.44 to 13.35]
Statistical Analysis 2: Comparison: MK-8457 100 mg BID vs Placebo; Treatment comparison of maxMAΔ in SBP from baseline to Day 10 after PM dosing; Test type: Superiority or Other; Linear mixed effects model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.94, 90% CI 2-sided [-5.68 to 3.81]
Statistical Analysis 3: Comparison: MK-8457 100 mg BID vs Placebo; Treatment comparison of maxMAΔ in DBP from baseline to Day 10 after AM dosing; Test type: Superiority or Other; Linear mixed effects model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.26, 90% CI 2-sided [0.81 to 9.71]
Statistical Analysis 4: Comparison: MK-8457 100 mg BID vs Placebo; Treatment comparison of maxMAΔ in DBP from baseline to Day 10 after PM dosing; Test type: Superiority or Other; Linear mixed effects model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.69, 90% CI 2-sided [-4.55 to 1.17]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours (AUC0-12hr) of MK-8457
Description: AUC0-12hr is an estimate of total plasma exposure to study drug over the dosing interval (12hr). Plasma concentrations of MK-8457 were determined on Day 1 (after initial dosing) and Day 10 (after multiple dosing). The placebo group is not included; this endpoint evaluated only the MK-8457 group.
Time Frame: pre-AM dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post AM dose on Days 1 and 10
Population: The per-protocol population consisting of participants who comply with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment according to the underlying scientific model used for analysis (AUC0-12hr).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | MK-8457 100 mg BID
Number analyzed (Participants) | 31
nM*hr
  Day 1 (n=31) | 29600 (36)
  Day 10 (n=30) | 56200 (44)

5. Secondary Outcome: Maximum Concentration (Cmax) of MK-8457
Description: Maximum plasma concentrations of MK-8521 were determined for the AM dose on Day 1 and Day 10. The placebo group was not included; this endpoint evaluated only the MK-8457 group.
Time Frame: pre-AM dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post AM dose on Days 1 and 10; 24 hrs post-AM dose on Day 10
Population: The per-protocol population consisting of participants who comply with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment according to the underlying scientific model used for analysis (Cmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-8457 100 mg BID
Number analyzed (Participants) | 31
nM
  Day 1 (n=31) | 5680 (31)
  Day 10 (n=30) | 8630 (38)

6. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8457
Description: Tmax was determined for the AM dose on Day 1 and Day 10. The placebo group was not included; this endpoint evaluated only the MK-8457 group.
Time Frame: as for outcome 5
Population: The per-protocol population consisting of participants who comply with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment according to the underlying scientific model used for analysis (Tmax).
Measure: Median (Full Range); unit: hr
Arm/Group | MK-8457 100 mg BID
Number analyzed (Participants) | 31
hr
  Day 1 (n=31) | 1 [0.75 to 2.0]
  Day 10 (n=30) | 1 [0.5 to 3.0]

7. Secondary Outcome: Trough Plasma Concentration (Ctrough) of MK-8457
Description: The lowest plasma concentration reached by the drug prior to the next administration was determined for Day 1 (after initial dosing) and Day 10 (after multiple dosing). The placebo group was not included; this endpoint evaluated only the MK-8457 group.
Time Frame: pre-AM dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hrs post AM dose on Days 1 and 10; pre-AM dose on Day 5 or 6
Population: The per-protocol population consisting of participants who comply with the protocol sufficiently to ensure that data were likely to exhibit the effects of treatment according to the underlying scientific model used for analysis (Ctrough).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-8457 100 mg BID
Number analyzed (Participants) | 31
nM
  Day 1 (n=31) | 999 (56)
  Day 10 (n=30) | 2540 (56)

8. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 70 days
Population: The safety population consisted of all participants who received at least one dose of the investigational drug.
Measure: Number; unit: Participant
Arm/Group | MK-8457 100 mg BID | Placebo
Number analyzed (Participants) | 31 | 29
Participant | 8 [-2.60 to 1.66] | 9 [-4.66 to -0.31]

9. Primary Outcome: Number of Participants Who Discontinued the Study Medication Due to an AE
Description: as for outcome 8
Time Frame: Up to 70 days
Population: The safety population consisted of all participants who received at least one dose of the investigational drug.
Measure: Number; unit: Participant
Arm/Group | MK-8457 100 mg BID | Placebo
Number analyzed (Participants) | 31 | 29
Participant | 1 [-2.60 to 1.66] | 0 [-4.66 to -0.31]

ADVERSE EVENTS:
Time Frame: Up to 70 days
Description: The safety population consisted of all participants who received at least one dose of the investigational drug.
Groups:
- MK-8457 100 mg BID: Participants received MK-8457 100 mg BID for 10 days
- Placebo: Participants received Placebo for MK-8457 for 10 days
Arm/Group | MK-8457 100 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 8/31 | 9/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8457 100 mg BID (N=31) | Placebo (N=29)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Energy decreased (General disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Swelling of fingers (General disorders) | 1 (1) | 0 (0)
Venipuncture site pain (General disorders) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
White blood cell count abnormal (Investigations) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.